CLINICAL TRIAL: NCT06137365
Title: A Randomized, Placebo-Controlled Clinical Trial of Once Daily Oral Cannabis for Weight Loss in Obese Individuals
Brief Title: Cannabis for Obesity Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Joshua A. Lile, Ph.D., Professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 86131
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: Placebo and active cannabis groups
Who Masked: Participant, Outcomes Assessor
Masking Description: Only investigator-level study personnel will have access to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Cannabis "gummy", starting at 2.5 mg THC and increased weekly by 2.5 mg increments up to a maximum target dose of 15 mg THC, administered once daily for duration of 6-month trial participation.
  Interventions: Drug: Cannabis
- Placebo (Placebo Comparator): Placebo cannabis "gummy", containing no active THC, administered once daily for duration of 6-month trial participation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabis — Cannabis gummy product will be prepared using cannabis flower extract.
  Arms: Active
Drug: Placebo — Placebo gummy product will be prepared using the same ingredients as the cannabis gummy but will not contain active cannabinoids.
  Arms: Placebo

SUMMARY:
The goal of this study is to determine the initial efficacy of once daily oral cannabis for weight loss in obese individuals.

ELIGIBILITY:
Inclusion Criteria

* Male or female.
* Age 18-65 years.
* BMI >=30 kg/m2 (i.e., obese).
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations at Screening and/or Check-in as assessed by one of the MD study personnel.
* Able to speak and read English.
* Apple or Android phone, or Android tablet with wi-fi or cellular service.
* Vital signs at Screening and Check-in as per the following ranges and stable (measured in a supine position after a minimum of 5 minutes of rest):

  * Systolic blood pressure ≥ 90 and ≤ 140 mmHg
  * Diastolic blood pressure ≥ 50 and ≤ 90 mmHg
  * Pulse rate ≥ 50 and ≤ 100 bpm

Exclusion Criteria

* Current cannabis use (e.g., past month; negative test for cannabinoids during screening) and no more than 15 self-reported lifetime uses.
* Self-reported current use of CBD.
* Severe past negative experience with cannabis or cannabinoid use (e.g., panic attack, anxiety).
* Use of any anti-obesity medication in the past 90 days. Specifically GLP-1 agonists (e.g., liraglutide, semaglutide, tirzepatide), SGLT-2 inhibitors (e.g., canagliflozin, dapagliflozin, empagliflozin, ertugliflozin), sulfonylureas (e.g., glimepiride, glipizide), medlitinides (e.g., repaglinide, nateglinide), Contrave, phentermine (alone or combination product such as Qsymia) or Orlistat. Stable use of metformin is permitted.
* Current treatment with insulin.
* History of type 1 diabetes.
* Stable body weight over the past 3 months. No changes greater than 5 kg.
* History of stomach or intestinal surgery or resection for obesity or otherwise (such as gastric bypass, sleeve-gastrectomy, bowel or small bowel resection) that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy, cholecystectomy, and hernia repair > 6 months prior to Screening will be allowed).
* Obesity secondary to a known genetic, endocrine, or medical condition, such as polycystic ovarian syndrome, hypothyroidism, Cushing's syndrome, growth hormone deficiency, insulinoma, hypothalamic disorders (e.g., Froelich syndrome, Bardet-Biedl syndrome, Prader-Willi syndrome)
* Moderate or Severe Substance Use Disorder according to DSM-5 criteria; urine test positive for recent use of an abused drug.
* History of significant psychiatric disorder (e.g., bipolar, schizophrenia, depression, history of panic attacks).
* Current use of psychiatric medications (e.g., antipsychotics, antidepressants, anxiolytics).
* Current or past year history of one or more of the following disorders associated with overeating: rumination disorder, bulimia nervosa, severe/extreme binge eating disorder (>7 episodes per week) or other specified/unspecified feeding/eating disorder that would increase risk to the participant or complicate interpretation of the data. Individuals who report mild to moderate (<7 episodes per week) binge eating disorder are eligible.
* Female participant who is pregnant, breast-feeding, or intends to become pregnant, or is of child-bearing potential and not using a highly effective contraceptive method.
* Any clinically important uncontrolled illness, medical/surgical procedure, or major trauma within 8 weeks prior to dose administration on Day 1.
* History of congestive heart failure or arrhythmias.
* Lab-Screening Exclusion:

  * Thyroid-stimulating hormone (TSH) level outside of the normal range, confirmed on repeat testing
  * AST, ALT, or alkaline phosphatase >2x ULN
  * EGFR <60 ml/min as calculated using the Cockroft-Gault equation.
* History of significant hypersensitivity, intolerance, or allergy to a cannabinoid or "gummy" product.
* Current use of any medications or supplement which would either compromise the validity of the study or the safety of the participant.
* History of seizure or predisposing factors for seizure (head trauma resulting in unconsciousness in past six months or CNS tumors).
* Any disorder, unwillingness, or inability, not covered by any of the other exclusion criteria, which in an investigator's opinion, might jeopardize the participant's safety or compliance with the protocol.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Weight change | weekly for duration of 6-month trial
  measured in kg using digital scale

IPD SHARING:
Plan to Share IPD: No